CLINICAL TRIAL: NCT04085016
Title: Effect of HMG-CoA Reductase Inhibitors on the Meibomian Gland Morphology in Patients With Meibomitis
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201610044RINB
Record Dates: First submitted 2019-09-08; First posted 2019-09-11 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Meibomian Gland Dysfunction; Meibomitis; Dyslipidemias
MeSH Terms: conditions — Meibomian Gland Dysfunction; Meibomitis; Dyslipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- meibography of statin group: patients with regular HMG CoA reductase inhibitor (statin) treatment
  Interventions: Device: Keratograph 5M, Oculus, Wetzlar, Germany
- meibography of non-statin group: patients with recently diagnosed dyslipidemia who were eligible to undergo 3 to 6 months of lifestyle interventions before re-evaluation for starting statin therapy
  Interventions: Device: Keratograph 5M, Oculus, Wetzlar, Germany

INTERVENTIONS:
Device: Keratograph 5M, Oculus, Wetzlar, Germany

SUMMARY:
This study intends to evaluate the relationship between meibomitis and statin use. Meibomitis is the predominant cause of evaporative dry eye. Higher cholesterol levels were noted in patients with meibomitis when compared to controls without meibomitis. We would like to investigate the effect of statin use on meibomitis among patients with dyslipidemia.

DETAILED DESCRIPTION:
The purpose of our study is to assess the change of meibomian gland structure in patients during treatment with 3-hydroxy-3-methyl-glutaryl-coenzyme A (HMG-CoA) reductase inhibitors using meibography. Patients with dyslipidemia with or without HMG-CoA reductase inhibitor (statin) treatment were recruited. Medical records are collected prospectively from Dec. 8th 2016 to Dec. 31st 2019. Meibomian gland (MG) morphology described by meiboscores, lid margin abnormality scores, meibum quality, and dry eye parameters were compared between the two groups. This study may also provide information about possible treatment options in patients with meibomitis in the future.

ELIGIBILITY:
Inclusion Criteria:

* patients with regular HMGCR inhibitor (statin) treatment, and those with recently diagnosed dyslipidemia who were eligible to undergo 3 to 6 months of lifestyle interventions before re-evaluation for starting statin therapy

Exclusion Criteria:

* patients with active eye infection, previous history of chemical or thermal injury to ocular surface, previous operation history of eyelid or conjunctiva, any known allergy or contraindications to statins, history of percutaneous coronary intervention, cerevascular accident, acute coronary syndrome, or rheumatological diseases, fish oil supplements or pregnancy were excluded

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with dyslipidemia
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2016-12-08 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
change in meiboscore | 6 months
  compare change in meibography images using meiboscore system

CONTACTS AND LOCATIONS:
Overall Officials: I-Jong Wang, MD,PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pinna A, Blasetti F, Zinellu A, Carru C, Solinas G. Meibomian gland dysfunction and hypercholesterolemia. Ophthalmology. 2013 Dec;120(12):2385-2389. doi: 10.1016/j.ophtha.2013.05.002. Epub 2013 Jun 6. PMID 23747164
- [Background] Nichols KK, Foulks GN, Bron AJ, Glasgow BJ, Dogru M, Tsubota K, Lemp MA, Sullivan DA. The international workshop on meibomian gland dysfunction: executive summary. Invest Ophthalmol Vis Sci. 2011 Mar 30;52(4):1922-9. doi: 10.1167/iovs.10-6997a. No abstract available. PMID 21450913
- [Background] Finis D, Ackermann P, Pischel N, Konig C, Hayajneh J, Borrelli M, Schrader S, Geerling G. Evaluation of Meibomian Gland Dysfunction and Local Distribution of Meibomian Gland Atrophy by Non-contact Infrared Meibography. Curr Eye Res. 2015;40(10):982-9. doi: 10.3109/02713683.2014.971929. Epub 2014 Oct 20. PMID 25330304